CLINICAL TRIAL: NCT00250289
Title: Invivo Study of the Efficacy of an Innovative Herbal Formula and Delivery System on Oral Malodor
Brief Title: Prevention of Oral Malodor With an Oral Sticker Containing Herbal Formula
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 191055HMO-CTIL
Record Dates: First submitted 2005-11-06; First posted 2005-11-08 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2009-10

CONDITIONS: Halitosis; Oral Malodor; Bad Breath
Keywords: malodor; halitosis; herbal formulation; natural medicinals; slow release delivery system
MeSH Terms: conditions — Halitosis

INTERVENTIONS:
Device: a mucosal sticker with herbal formula

SUMMARY:
the use of a herbal formulation containing sage, echinacea,lavender and mastic gum would prevent oral malodor if delivered in an appropriate delivery system to enable slow release of the active ingredients.

DETAILED DESCRIPTION:
Oral malodor (Halitosis, Fetor ex ora) is a common and disturbing condition, affecting according to some studies about one quarter of the population. This condition may start at any time from early childhood through adolescence, adulthood and old age and vary in character and severity.The bacteria responsible for malodor production are for the most part Gram negative oral bacteria (2- 4) such as Porphyromonas gingivalis, Fusobacterium nucleatum and Prevotella intermedia. These bacteria reside on various locations within the oral cavity (e.g. tongue dorsum, interdental space, periodontal pockets, tonsils) and breakdown salivary and oral proteins into their amino acid building blocks. Some of these amino acids (e.g. methionine, cysteine, tryptophan, lysine) are further metabolized yielding malodorous volatile products such as methylmercaptan, hydrogen sulfide, indole, skatole and cadaverine (5-7). These are foul smelling compounds, which are released during exhalation and speech.in our study we intend to use an aprooved mucosal sticker containing carbopol and hydroxypropylcellulose mixed with the herbal ingredients and placed on the palatal mucosa.than mesure the volatile sulfur compounds to observe if the composition has antimalodor effect and for how long. the herbal ingredients are used for many years for medicinal and nutritional purposes. if our hypothesis is right we might have another formulation and method of application to prevent oral malodor

ELIGIBILITY:
Inclusion Criteria:

* random gender, age and healthy people

Exclusion Criteria:

* used antibiotics in the last three months or suffer from systemic disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-01 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Oral malodor will be measured with a Halimeter monitor and an odor judge before the sticker application and following the application every 7 minutes until the odor level would reach plateau.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Perez Davidi, DMD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel

REFERENCES:
- [Result] Mizrahi B, Golenser J, Wolnerman JS, Domb AJ. Adhesive tablet effective for treating canker sores in humans. J Pharm Sci. 2004 Dec;93(12):2927-35. doi: 10.1002/jps.20193. PMID 15459950
- See also: Michael Perez Davidi — http://www.mypd.co.il